CLINICAL TRIAL: NCT01142908
Title: Cardiovascular Intervention Improvement Telemedicine Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 08-297; 08-297 (Other Grant/Funding Number: VA HSRD)
Record Dates: First submitted 2010-05-24; First posted 2010-06-11 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Disease; Hypertension; Diabetes; Hyperlipidemia
Keywords: Cardiovascular Disease; Hypertension; Diabetes; Hyperlipidemia; Adherence
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): The pharmacist CVD intervention group - clinical pharmacist-administered intervention which focuses on behavioral and medication management for 12 months.
  Interventions: Behavioral: Pharmacist CVD
- Arm 2 (No Intervention): The education control group - these participants will receive educational material about CVD reduction.

INTERVENTIONS:
Behavioral: Pharmacist CVD — clinical pharmacist-administered intervention which focuses on behavioral and medication management for 12 months.
  Arms: Arm 1

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the United States; more than 80% of veterans have > 2 risk factors for CVD. Our study is one of the first to examine the implementation of a tailored behavioral/educational self-management intervention in primary care clinics designed to improve CVD risk. The proposed study could result in a leap forward in CVD risk management among veterans for several reasons: 1) ) This is a novel extension of our previous interventions that have demonstrated improved BP, now designed to address multiple chronic conditions contributing to CVD risk, particularly hyperlipidemia and diabetes. The study focuses on both multiple CVD-related risk factor management and medication management 2) The intervention is multi-behavioral; it addresses patients' various health behavior (e.g., smoking, diet, and medication adherence). 3) Components of the intervention will include specific recommendations and transportability of intervention application software and tracking packages that will allow clinic managers to implement the intervention if it is effective.

DETAILED DESCRIPTION:
Anticipated Impacts on Veteran's Healthcare: Cardiovascular disease (CVD) is the leading cause of death in the U.S.; more than 80% of veterans have > 2 risk factors for CVD. An intervention that addresses multiple CVD risk factors among high-risk veterans has the greatest potential to improve morbidity and mortality.

Project Background/Rationale: The proposed study will take place in two VA primary care clinics (1-Community-Based Outpatient Clinics and 1-primary care clinic affiliated with a hospital). We will improve CVD risk among veterans by addressing the modifiable risk factors of systolic blood pressure (SBP), smoking, and low-density lipoprotein cholesterol (LDL-C). The intervention will be tailored to the needs of vulnerable high risk patients (e.g. African Americans, low literate) and integrated into clinics, thereby enhancing the potential for benefit and generalizability to other settings.

The proposed study could significantly improve CVD risk management among veterans for several reasons: 1) This intervention is a novel extension of our previous efficacious interventions, but provides a novel extension to address multiple chronic conditions contributing to CVD risk. 2) The intervention focuses on both multiple CVD-related behaviors and medication management. 3) The intervention was developed to ensure implementation across a large and representative sample of veterans; and; 4) The intervention, if found efficacious and financially self-sustaining, could be widely implemented within the VA healthcare system.

Project Objectives: The proposed study will examine two research questions:

1. Can patients randomized to a clinical pharmacist-administered telephone behavioral/ medication management intervention tailored to their needs improve CVD outcomes relative to a control group over 12 months? Primary Hypothesis: (H1) Veterans who receive the behavioral/medication intervention will have greater improvement of their CVD Risk Profile over the 12 months of follow-up as compared to the control group.

   Secondary Hypotheses: (H2) Veterans who receive the intervention will have improved medication adherence, physical activity, improved diet, lower body mass index as compared to the control group over 12 months of follow-up. (H3) Veterans who receive the intervention will have greater improvements in LDL over the 12 months of follow-up as compared to the control group. (H4) Veterans with diabetes who receive the intervention will have greater improved HbA1c as compared to the control group over 12 months of follow-up.
2. If the intervention is found to be effective, is it cost effective? Project Methods: To address these hypotheses, we propose a two-arm randomized clinical trial design in which 500 patients with cardiovascular disease will be randomized to either the education control group or the intervention group. Patients randomized to the intervention group will receive a clinical pharmacist-administered intervention, which focuses on behavioral and a medication management. The intervention will occur over 12 months. Patients randomized to the control group will receive educational material about CVD reduction. Given the national prevalence of CVD and the dismal rates of risk factor control, intensive, but easily disseminated interventions such as the one proposed could significantly improve treatment of this epidemic in the VA.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in one of three Durham Veterans Affairs Medical Center (DVAMC) Primary Care Clinics affiliated with the hospital or the Raleigh Community-Based Outpatient Clinic (CBOC) for at least one year;
* At least one visit to a primary care physician (PCP) at the Raleigh CBOC or Durham Veterans Affairs Medical Center (VAMC) associated primary care clinics in the previous 12 months;
* Outpatient diagnostic code for hypertension and/or hypercholesterolemia and lab values indicating either poorly controlled BP levels (>150/90 Hg) AND/OR LDL (>130mg/dl) in the previous year.

Exclusion Criteria:

* diagnosed with metastatic cancer,
* diagnosed with dementia,
* active diagnosis of psychosis,
* treated with dialysis,
* most recent creatinine lab level >2.5 or no creatinine lab value within past year
* hospitalized for a stroke, heart attack, or had surgery for blocked arteries in the past 3 months,
* participating in another interventional trial,
* not currently receiving care at the Durham VAMC or the Raleigh CBOC
* resident of a nursing home,
* hard time seeing type/printing on books, magazines articles, etc.
* hard time hearing on the telephone
* limited/no access to telephone
* plans to move medical care from DVAMC or Raleigh CBOC in next 12 months
* CVD care is currently being managed by a clinical pharmacist
* HbA1C value in the last 90day > 10% and patient is currently not on an insulin regimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B Bosworth, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goldstein KM, Stechuchak KM, Zullig LL, Oddone EZ, Olsen MK, McCant FA, Bastian LA, Batch BC, Bosworth HB. Impact of Gender on Satisfaction and Confidence in Cholesterol Control Among Veterans at Risk for Cardiovascular Disease. J Womens Health (Larchmt). 2017 Jul;26(7):806-814. doi: 10.1089/jwh.2016.5739. Epub 2017 Feb 13. PMID 28192012
- [Result] Goldstein KM, Oddone EZ, Bastian LA, Olsen MK, Batch BC, Washington DL. Characteristics and Health Care Preferences Associated with Cardiovascular Disease Risk among Women Veterans. Womens Health Issues. 2017 Nov-Dec;27(6):700-706. doi: 10.1016/j.whi.2017.08.002. Epub 2017 Sep 8. PMID 28890128
- [Result] Bosworth HB, Olsen MK, McCant F, Stechuchak KM, Danus S, Crowley MJ, Goldstein KM, Zullig LL, Oddone EZ. Telemedicine cardiovascular risk reduction in veterans: The CITIES trial. Am Heart J. 2018 May;199:122-129. doi: 10.1016/j.ahj.2018.02.002. Epub 2018 Feb 10. PMID 29754649
- [Result] Melnyk SD, Zullig LL, McCant F, Danus S, Oddone E, Bastian L, Olsen M, Stechuchak KM, Edelman D, Rakley S, Morey M, Bosworth HB. Telemedicine cardiovascular risk reduction in veterans. Am Heart J. 2013 Apr;165(4):501-8. doi: 10.1016/j.ahj.2012.08.005. Epub 2013 Feb 28. PMID 23537965
- [Result] Zullig LL, Melnyk SD, Stechuchak KM, McCant F, Danus S, Oddone E, Bastian L, Olsen M, Edelman D, Rakley S, Morey M, Bosworth HB. The Cardiovascular Intervention Improvement Telemedicine Study (CITIES): rationale for a tailored behavioral and educational pharmacist-administered intervention for achieving cardiovascular disease risk reduction. Telemed J E Health. 2014 Feb;20(2):135-43. doi: 10.1089/tmj.2013.0145. Epub 2013 Dec 4. PMID 24303930
- [Result] Zullig LL, Stechuchak KM, Goldstein KM, Olsen MK, McCant FM, Danus S, Crowley MJ, Oddone EZ, Bosworth HB. Patient-reported medication adherence barriers among patients with cardiovascular risk factors. J Manag Care Spec Pharm. 2015 Jun;21(6):479-85. doi: 10.18553/jmcp.2015.21.6.479. PMID 26011549
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Ulmer CS, McCant F, Stechuchak KM, Olsen M, Bosworth HB. Prevalence of insomnia disorder and sleep apnea in a sample of veterans at risk for cardiovascular disease. J Clin Sleep Med. 2021 Jul 1;17(7):1441-1446. doi: 10.5664/jcsm.9228. PMID 33688827
- [Derived] Zullig LL, Oakes MM, McCant F, Bosworth HB. Lessons learned from two randomized controlled trials: CITIES and STOP-DKD. Contemp Clin Trials Commun. 2020 Jul 8;19:100612. doi: 10.1016/j.conctc.2020.100612. eCollection 2020 Sep. PMID 32685766
- [Derived] Goldstein KM, Melnyk SD, Zullig LL, Stechuchak KM, Oddone E, Bastian LA, Rakley S, Olsen MK, Bosworth HB. Heart matters: Gender and racial differences cardiovascular disease risk factor control among veterans. Womens Health Issues. 2014 Sep-Oct;24(5):477-83. doi: 10.1016/j.whi.2014.05.005. PMID 25213741

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacist CVD: The pharmacist cardiovascular (CVD) intervention group - clinical pharmacist-administered intervention which focuses on behavioral and medication management for 12 months.
- Education Control: The education control group - these participants will receive educational material about CVD reduction.
Period: Overall Study
Arm/Group | Pharmacist CVD | Education Control
Started | 215 | 213
6 Month f/u | 188 | 196
Completed | 183 | 191
Not Completed | 32 | 22
Not completed — Lost to Follow-up | 19 | 13
Not completed — Death | 1 | 4
Not completed — Excluded - did not meet criteria | 9 | 5
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pharmacist CVD: The pharmacist CVD intervention group - clinical pharmacist-administered intervention which focuses on behavioral and medication management for 12 months.
- Total: Total of all reporting groups
Arm/Group | Pharmacist CVD | Education Control | Total
Number analyzed (Participants) | 215 | 213 | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.4) | 61.5 (8.9) | 61.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 182 | 181 | 363
Race/Ethnicity, Customized [Number; unit: participants]
  White | 93 | 106 | 199
  Black | 111 | 102 | 213
  Other | 10 | 4 | 14
  Refused/Missing | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 215 | 213 | 428

OUTCOME MEASURES:

1. Primary Outcome: Framingham Risk Percent (Estimate of 10 Year Risk of Cardiovascular Disease in Percent)
Description: Components of the Framingham include gender, age fixed at baseline, systolic blood pressure (presence/absence of blood pressure medications at each time point [combination of administrative med data pull and self-report at assessment]), total cholesterol, HDL cholesterol, smoking status (assessed via self-report at each study survey), and diabetes (diabetes is a combination of self-report and VA Computerized Patient Record System (CPRS) data review). "New cases" of diabetes are allowed to be updated at 6 and 12 months f/u.
Time Frame: Baseline
Population: Two out of the 215 participants in the Pharmacist CVD group had missing data due to not having the blood pressure component of the Framingham collected at baseline.
Measure: Mean (Standard Deviation); unit: % 10 yr Risk
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 213 | 213
% 10 yr Risk | 32.4 (18.8) | 31.6 (18.6)

2. Secondary Outcome: Mean Systolic Blood Pressure
Description: Mean BP is calculated as the average of 3 bp measurements. Collected during BP outcome measurement conducted at interviews
Time Frame: Baseline
Population: One out of the 215 participants in the Pharmacist CVD group did not have blood pressure collected at baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 214 | 213
mmHg | 130.6 (18.5) | 129.7 (18.8)

3. Secondary Outcome: Mean Systolic Blood Pressure
Description: as for outcome 2
Time Frame: 6 months
Population: 28 out of the 215 participants in the Pharmacist CVD group and 23 out of the 213 in the Education Control group had missing blood pressure measurement at 6 months due to missing the 6 month interview entirely or blood pressure not collected at the 6 month assessment due to patient arm size exceeding cuff size or interview completed over the phone.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 187 | 190
mmHg | 128.3 (16.5) | 127.7 (16.8)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 6 months; Test type: Superiority or Other; p = 0.93, Mixed Models Analysis; Adjusted for gender, diabetes, and smoking status stratification variables; Mean Difference (Net) = 0.1, 95% CI 2-sided [-2.8 to 3.1] — Direction of the test of comparison is Pharmacist Intervention minus Control

4. Secondary Outcome: Mean Systolic Blood Pressure
Description: as for outcome 2
Time Frame: 12 months
Population: 36 out of the 215 participants in the Pharmacist CVD group and 30 out of the 213 in the Education Control group had missing blood pressure measurement at 12 mo. due to missing the 12 month interview entirely or blood pressure not collected at the 12 month assessment due to patient arm size exceeding cuff size or interview completed over the phone.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 179 | 183
mmHg | 128.5 (15.4) | 126.4 (16.2)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 12 months; Test type: Superiority or Other; p = 0.34, Mixed Models Analysis; Adjusted for gender, diabetes, and smoking status stratification variables; Mean Difference (Net) = 1.4, 95% CI 2-sided [-1.5 to 4.3] — Direction of the test of comparison is Pharmacist Intervention minus Control

5. Secondary Outcome: Mean Diastolic Blood Pressure
Description: as for outcome 2
Time Frame: Baseline
Population: One out of the 215 participants in the Pharmacist CVD group did not have blood pressure collected at baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 214 | 213
mmHg | 75.8 (11.5) | 75.8 (12.4)

6. Secondary Outcome: Mean Diastolic Blood Pressure
Description: as for outcome 2
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 187 | 190
mmHg | 74.0 (11.0) | 74.1 (11.9)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 6 months; Test type: Superiority or Other; p = 0.91, Mixed Models Analysis; Adjusted for gender, diabetes, and smoking status stratification variables; Mean Difference (Net) = -0.1, 95% CI 2-sided [-2.0 to 1.8] — Direction of the test of comparison is Pharmacist Intervention minus Control

7. Secondary Outcome: Mean Diastolic Blood Pressure
Description: as for outcome 2
Time Frame: 12 months
Population: 36 out of the 215 participants in the Pharmacist CVD group and 30 out of the 213 in the Education Control group had missing blood pressure measurement at 12 months due to missing the 12 month interview entirely or blood pressure not collected at the 12 mo. assessment due to patient arm size exceeding cuff size or interview completed over the phone.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 179 | 183
mmHg | 73.4 (10.3) | 73.1 (10.9)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 12 months; Test type: Superiority or Other; p = 0.70, Mixed Models Analysis; Adjusted for gender, diabetes, and smoking status stratification variables; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.5 to 2.2] — Direction of the test of comparison is Pharmacist Intervention minus Control

8. Primary Outcome: Framingham Risk Percent (Estimate of 10 Year Risk of Cardiovascular Disease in Percent)
Description: Components of the Framingham include gender, age fixed at baseline, systolic blood pressure (presence/absence of blood pressure medications at each time point [combination of administrative med data pull and self-report at assessment]), total cholesterol, HDL cholesterol, smoking status (assessed via self-report at each study survey), and diabetes (diabetes is a combination of self-report and CPRS data review). "New cases" of diabetes are allowed to be updated at 6 and 12 months f/u.
Time Frame: 6 months
Population: 29 out of the 215 participants in the Pharmacist CVD group and 24 of the 213 participants in the Education Control group had missing data at 6 months due to entirely missing the 6 month assessment or having missing data on one or more of the Framingham components.
Measure: Mean (Standard Deviation); unit: % 10 yr Risk
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 186 | 189
% 10 yr Risk | 30.0 (17.2) | 30.2 (18.7)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 6 months; Test type: Superiority or Other; p = 0.1, Mixed Models Analysis; Mean Difference (Net) = -1.8, 95% CI 2-sided [-3.9 to 0.3] — Direction of the test of comparison is Pharmacist Intervention minus Control

9. Primary Outcome: Framingham Risk Percent (Estimate of 10 Year Risk of Cardiovascular Disease in Percent)
Description: as for outcome 8
Time Frame: 12 months
Population: 43 out of the 215 participants in the Pharmacist CVD group and 33 of the 213 participants in the Education Control group had missing data at 12 months due to entirely missing the 12 month assessment or having missing data on one or more of the Framingham components.
Measure: Mean (Standard Deviation); unit: % 10 yr Risk
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 172 | 180
% 10 yr Risk | 28.9 (15.5) | 28.4 (18.3)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 12 months; Test type: Superiority or Other; p = 0.74, Mixed Models Analysis; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.4 to 1.7] — Direction of the test of comparison is Pharmacist Intervention minus Control

10. Secondary Outcome: Medication Non-adherence
Description: First 4 items of the 5 item Morisky Self-reported measure of medication adherence was used to determine medication non-adherence.
Time Frame: Baseline
Population: 5 out of the 215 participants in the Pharmacist CVD group and 2 out of the 213 participants in the Education Control group had missing data for medication non-adherence due to non-response of adherence items collected in the baseline interview.
Measure: Number; unit: participants
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 210 | 211
participants | 137 | 110

11. Secondary Outcome: Medication Non-adherence
Description: as for outcome 10
Time Frame: 6 months
Population: 28 out of the 215 participants in the Pharmacist CVD group and 18 out of the 213 participants in the Education Control group had missing data for medication non-adherence due to missing the 6 month assessment or non-response of adherence items collected in the 6 month interview.
Measure: Number; unit: participants
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 187 | 195
participants | 92 | 85
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 6 months; Test type: Superiority or Other; p = 0.87, Gen. Est. Equation with a Logit Link; Method Used Expanded: Generalized Estimating Equation with a Logit Link. Adjusted for gender, diabetes, and smoking status stratification variables; logit-difference (Net) = -0.03, 95% CI 2-sided [-0.4 to 0.3] — Direction of the test of comparison is Pharmacist Intervention minus Control

12. Secondary Outcome: Medication Non-adherence
Description: as for outcome 10
Time Frame: 12 months
Population: 35 out of the 215 participants in the Pharmacist CVD group and 24 out of the 213 participants in the Education Control group had missing data for medication non-adherence due to missing the 12 month assessment or non-response of adherence items collected in the 12 month interview.
Measure: Number; unit: participants
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 180 | 189
participants | 96 | 82
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 12 months; Test type: Superiority or Other; p = 0.36, Gen. Est. Equation with a Logit Link; [statistical method as in outcome 11, analysis 1]; logit-difference (Net) = 0.2, 95% CI 2-sided [-0.2 to 0.5] — Direction of the test of comparison is Pharmacist Intervention minus Control

13. Secondary Outcome: Cholesterol LDL
Description: Collected during interview visit by lab personnel
Time Frame: Baseline
Population: 4 out of the 215 participants in the Pharmacist CVD group and 2 out of the 213 participants in the Education Control group had missing data due to not having cholesterol LDL collected at baseline.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 211 | 211
mg/dL | 125.5 (37.3) | 123.9 (36.2)

14. Secondary Outcome: Cholesterol LDL
Description: Collected during interview visit by lab personnel
Time Frame: 6 months
Population: 29 out of the 215 participants in the Pharmacist CVD group and 22 out of the 213 in the Education Control group had missing cholesterol LDL at 6 months due to missing the 6 month interview entirely or not completing the lab assessment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 186 | 191
mg/dL | 114.9 (34.9) | 118.9 (34.3)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 6 months; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis; Adjusted for gender, diabetes, and smoking status stratification variables; Mean Difference (Net) = -4.9, 95% CI 2-sided [-10.3 to 0.6] — Direction of the test of comparison is Pharmacist Intervention minus Control

15. Secondary Outcome: Cholesterol LDL
Description: Collected during interview visit by lab personnel
Time Frame: 12 months
Population: 34 out of the 215 participants in the Pharmacist CVD group and 27 out of the 213 in the Education Control group had missing cholesterol LDL at 12 months due to missing the 12 month interview entirely or not completing the lab assessment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 181 | 186
mg/dL | 114.4 (36.8) | 115.3 (34.0)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 12 months; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis; Adjusted for gender, diabetes, and smoking status stratification variables; Mean Difference (Net) = -0.8, 95% CI 2-sided [-6.6 to 5.0] — Direction of the test of comparison is Pharmacist Intervention minus Control

16. Secondary Outcome: Body Mass Index
Description: Calculated from vitals (height & weight) obtained during interview
Time Frame: Baseline
Population: 5 out of the 215 participants in the Pharmacist CVD group and 1 out of the 213 participants in the Education Control group had missing data due weight and/or height not collected at baseline.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 210 | 212
kg/m^2 | 31.9 (5.8) | 31.6 (5.7)

17. Secondary Outcome: Body Mass Index
Description: Calculated from vitals (height & weight) obtained during interview
Time Frame: 6 months
Population: 30 out of the 215 participants in the Pharmacist CVD group and 23 out of the 213 in the Education Control group had missing body mass index at 6 months due to missing the 6 month interview entirely or the interview was completed over the phone, or weight was not obtained at the 6 month interview.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 185 | 190
kg/m^2 | 32.1 (6.3) | 31.5 (5.4)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 6 months; Test type: Superiority or Other; p = 0.83, Mixed Models Analysis; Adjusted for gender, diabetes, and smoking status stratification variables; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.2 to 0.2] — Direction of the test of comparison is Pharmacist Intervention minus Control

18. Secondary Outcome: Body Mass Index
Description: Calculated from vitals (height & weight) obtained during interview
Time Frame: 12 months
Population: 39 out of the 215 participants in the Pharmacist CVD group and 31 out of the 213 in the Education Control group had missing body mass index at 12 months due to missing the 12 month interview entirely or the interview was completed over the phone, or weight was not obtained at the 12 month interview.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 176 | 182
kg/m^2 | 31.9 (6.0) | 31.6 (5.7)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 12 months; Test type: Superiority or Other; p = 0.54, Mixed Models Analysis; Adjusted for gender, diabetes, and smoking status stratification variables; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.2] — Direction of the test of comparison is Pharmacist Intervention minus Control

19. Secondary Outcome: HBA1C in Diabetic Patients
Description: Lab values collected at interview visit by lab personnel
Time Frame: Baseline
Population: 4 out of the 85 participants in the Pharmacist CVD group with diabetes at baseline and 2 out of the 86 participants in the Education Control group with diabetes at baseline had missing data due to not having HBA1C collected at baseline.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 81 | 84
percentage of glycosylated hemoglobin | 8.0 (2.3) | 7.6 (1.7)

20. Secondary Outcome: HBA1C in Diabetic Patients
Description: Lab values collected at interview visit by lab personnel
Time Frame: 6 months
Population: 12 out of the 85 participants in the Pharmacist CVD group with diabetes at baseline and 11 out of the 86 participants in the Education Control group with diabetes at baseline had missing HBA1C at 6 months due to missing the 6 month interview entirely or not completing the lab assessment.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 73 | 75
percentage of glycosylated hemoglobin | 7.5 (1.8) | 7.7 (1.8)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 6 months; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis; Adjusted for gender and smoking status stratification variables; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.2] — Direction of the test of comparison is Pharmacist Intervention minus Control

21. Secondary Outcome: HBA1C in Diabetic Patients
Description: Lab values collected at interview visit by lab personnel
Time Frame: 12 months
Population: 14 out of the 85 participants in the Pharmacist CVD group with diabetes at baseline and 15 out of the 86 participants in the Education Control group with diabetes at baseline had missing HBA1C at 6 months due to missing the 6 month interview entirely or not completing the lab assessment.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Pharmacist CVD | Education Control
Number analyzed (Participants) | 71 | 71
percentage of glycosylated hemoglobin | 7.5 (1.8) | 7.7 (1.7)
Statistical Analysis 1: Comparison: Pharmacist CVD vs Education Control; Comparison at 12 months; Test type: Superiority or Other; p = 0.72, Mixed Models Analysis; Adjusted for gender and smoking status stratification variables; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.4] — Direction of the test of comparison is Pharmacist Intervention minus Control

ADVERSE EVENTS:
Time Frame: Adverse events were collected through out the study from baseline thru completion.
Description: Adverse events information was collected by questionnaire from patients at 6 month and 12 month outcome assessments. Adverse event information was also collected from patients through contact with the Pharmacist interventionist or if during updating of clinical records it was discovered that an adverse event had occurred with a patient.
Arm/Group | Pharmacist CVD | Education Control
Serious Adverse Events (participants affected / at risk) | 126/215 | 123/213
Other Adverse Events (participants affected / at risk) | 0/215 | 0/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacist CVD (N=215) | Education Control (N=213)
Non_Cardiac Pain (Blood and lymphatic system disorders) | 1 (2) | 0
Emergecy Room Visit (Blood and lymphatic system disorders) | 2 (2) | 0
Coronary Issues (Cardiac disorders) | 3 (4) | 7 (8)
Emergency room visit (Cardiac disorders) | 21 (34) | 15 (15)
Non_Cardiac Pain (Cardiac disorders) | 2 (2) | 0
Orthopedic (Cardiac disorders) | 1 (1) | 0
Planned Surgery (Cardiac disorders) | 0 | 2 (2)
Study Safety Protocol (Cardiac disorders) | 10 (10) | 13 (16)
Emergency room visit (Ear and labyrinth disorders) | 3 (3) | 4 (6)
Infection (Ear and labyrinth disorders) | 0 | 1 (1)
Non_Cardiac Pain (Ear and labyrinth disorders) | 1 (1) | 0
Death (Endocrine disorders) | 0 | 1 (1)
Emergency room visit (Endocrine disorders) | 4 (7) | 9 (13)
Endocrine (Endocrine disorders) | 2 (2) | 1 (1)
Non_Cardiac Pain (Endocrine disorders) | 1 (1) | 0
Emergency room visit (Eye disorders) | 1 (1) | 5 (6)
Optometry (Eye disorders) | 0 | 2 (3)
Planned Surgery (Eye disorders) | 0 | 1 (1)
Emergency room visit (Gastrointestinal disorders) | 18 (21) | 13 (16)
Gastro_Intestinal (Gastrointestinal disorders) | 0 | 1 (1)
Planned Surgery (Gastrointestinal disorders) | 0 | 1 (1)
Allergic Reaction (non_med SE) (General disorders) | 1 (1) | 0
Death (General disorders) | 0 | 2 (2)
Emergency room visit (General disorders) | 14 (23) | 21 (22)
Medication Refill (General disorders) | 1 (1) | 1 (1)
Neurologic (General disorders) | 1 (2) | 0
Non_Cardiac Pain (General disorders) | 2 (2) | 2 (4)
Planned Surgery (General disorders) | 2 (2) | 0
Psychological (General disorders) | 1 (1) | 0
Emergency room visit (Infections and infestations) | 22 (22) | 5 (6)
Gastro_Intestinal (Infections and infestations) | 0 | 1 (1)
Infection (Infections and infestations) | 6 (8) | 2 (2)
Medication Refill (Infections and infestations) | 0 | 1 (1)
Emergency room visit (Injury, poisoning and procedural complications) | 3 (4) | 1 (3)
Non_Cardiac Pain (Injury, poisoning and procedural complications) | 1 (1) | 0
Protocol Deviation (Investigations) | 2 (2) | 0
Study Safety Protocol (Investigations) | 2 (2) | 0
Emergency room visit (Metabolism and nutrition disorders) | 1 (1) | 0
Circulatory (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Emergency room visit (Musculoskeletal and connective tissue disorders) | 27 (37) | 30 (44)
Endocrine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Neurologic (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Non_Cardiac Pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 3 (3)
Orthopedic (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Dermatologic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Emergency room visit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Protocol Deviation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Coronary issues (Nervous system disorders) | 0 | 1 (1)
Emergency room visit (Nervous system disorders) | 2 (2) | 2 (2)
Neurologic (Nervous system disorders) | 1 (1) | 3 (3)
Non_Cardiac Pain (Nervous system disorders) | 1 (1) | 0
Emergency room visit (Psychiatric disorders) | 5 (7) | 5 (5)
Medication Refill (Psychiatric disorders) | 1 (1) | 0
Non_Cardiac Pain (Psychiatric disorders) | 1 (2) | 0
Psychological (Psychiatric disorders) | 4 (4) | 4 (4)
Emergency room visit (Renal and urinary disorders) | 4 (5) | 5 (5)
Endocrine (Renal and urinary disorders) | 1 (1) | 0
Non_Cardiac Pain (Renal and urinary disorders) | 1 (1) | 0
Planned Surgery (Renal and urinary disorders) | 1 (1) | 0
Non_Cardiac Pain (Reproductive system and breast disorders) | 0 | 1 (1)
Emergency room visit (Reproductive system and breast disorders) | 3 (4) | 0
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Emergency room visit (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 12 (14)
Infection (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Dermatologic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Emergency room visit (Skin and subcutaneous tissue disorders) | 5 (7) | 6 (8)
Infection (Skin and subcutaneous tissue disorders) | 0 | 3 (3)
Emergency room visit (Social circumstances) | 0 | 1 (1)
Coronary issues (Surgical and medical procedures) | 1 (1) | 1 (1)
Emergency room visit (Surgical and medical procedures) | 2 (2) | 1 (2)
Gastro_Intestinal (Surgical and medical procedures) | 0 | 1 (1)
Infection (Surgical and medical procedures) | 0 | 1 (1)
Orthopedic (Surgical and medical procedures) | 3 (3) | 1 (1)
Planned Surgery (Surgical and medical procedures) | 18 (19) | 9 (10)
Pulmonary (Surgical and medical procedures) | 1 (1) | 0
Circulatory (Vascular disorders) | 1 (1) | 0
Coronary issues (Vascular disorders) | 1 (1) | 1 (1)
Emergency room visit (Vascular disorders) | 1 (2) | 3 (3)
Neurologic (Vascular disorders) | 1 (1) | 1 (1)
Planned Surgery (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes